CLINICAL TRIAL: NCT01002599
Title: Does BoussignacTM CPAP Compared to Venturi Mask Improve Oxygenation and Pulmonary Function in Morbidly Obese Patients Undergoing Bariatric Surgery?
Brief Title: Oxygenation and Pulmonary Function in Morbidly Obese Patients Undergoing Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. David Wong, University Health Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-0160-B
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Morbid Obesity
Keywords: bariatric surgery; morbidly obese; BMI >35; CPAP; Venturi; Boussignac; Ventilation; Pulmonary function; Morbidly Obese Patients undergoing bariatric surgery
MeSH Terms: conditions — Obesity, Morbid; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Boussignac TM CPAP (Experimental): Post-operative patients will be fitted with a Boussignac TM CPAP mask immediately after extubation and oxygenation and pulmonary function will be measured over a 24 hour period.
  Interventions: Device: Boussignac TM CPAP
- Venturi Face Mask (Active Comparator): Post-operative patients will be fitted with a Venturi face mask immediately after extubation and oxygenation and pulmonary function will be measured over a 24 hour period.
  Interventions: Device: Venturi Face Mask

INTERVENTIONS:
Device: Boussignac TM CPAP — Post-operative patients will be fitted with a Boussignac TM CPAP mask immediately after extubation and oxygenation and pulmonary function will be measured over a 24 hour period.
  Arms: Boussignac TM CPAP
Device: Venturi Face Mask — Post-operative patients will be fitted with a Venturi face mask immediately after extubation and oxygenation and pulmonary function will be measured over a 24 hour period.
  Arms: Venturi Face Mask

SUMMARY:
This is a randomized controlled study in which morbidly obese patients undergoing bariatric surgery will be recruited in the preoperative clinic. Patients will be randomized into 2 groups to receive oxygen with Boussignac TM continuous positive airway pressure (CPAP) or conventional Venturi mask postoperatively immediately after extubation. The objective of the study is to examine if Boussignac TM CPAP results in improved oxygenation versus Venturi face mask when it is applied immediately after extubation in morbidly obese patients post bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 18 to 75 years of age
* American Society of Anesthesiologists' (ASA) class I to III
* Morbidly obese with a body mass index > 35 kg/m2
* Patients undergoing bariatric surgery

Exclusion Criteria:

* Patient refusal
* Pre-existing cardiac failure, asthma, chronic obstructive pulmonary disease or interstitial pulmonary disease
* Systolic blood pressure less than 90 mmHg despite pharmacotherapy
* Hb < 70 g/L
* Impaired gastric emptying
* Severe psychiatric disorder
* Language barrier

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio (PF ratio) immediately on arrival to postanesthesia care unit, 1 hour, 2 hours, and 24 hours post-extubation. | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada